CLINICAL TRIAL: NCT03774264
Title: Treatment Response to Xiaflex Based on Ultrasound Characterization of Plaque for Men With Peyronie's Disease
Brief Title: Treatment Response to Xiaflex for Men With Peyronie's Disease
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: Endo Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Ranjith Ramasamy, MD, Director of Male Fertility and Andrology, University of Miami, University of Miami
Other Study IDs: 20180188
Record Dates: First submitted 2018-12-03; First posted 2018-12-12 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Peyronie Disease
MeSH Terms: conditions — Penile Induration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Xiaflex group: Patients will be evaluated in our urology clinic at baseline for possible inclusion in our study. All patients at baseline evaluation will be evaluated for duration of symptoms, relationship stability, IIEF and PDQ. All patients will obtain a penile Doppler ultrasound with the aid of a vasoactive substance by a specially trained technician. During this visit, plaque measurements will be taken: location of plaque, distance of plaque from the tip of the penis, degree of curvature measured by goniometer.
  Ultrasound characteristics will be documented: Type (Type 1: The plaque appears as a thickening of the tunica albuginea without acoustic shadowing. Type 2: A moderately calcified plaque with a typical ultrasound shadow. Type 3: A severely calcified plaque with typical ultrasound shadowing) and Grade of calcification (grade 1 (<0.3 cm), grade 2 (>0.3 cm, <1.5 cm), grade 3 (>1.5 cm; or ≥ 2 plaques >1.0 cm). Sample data sheet attached as appendix 2.

SUMMARY:
The purpose of this research study is to develop a database of patients with Peyronie's disease who are treated at the University of Miami. The collected data will help the researchers to better understand Peyronie's disease and its response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Able to provide informed consent
* A stable relationship for ≥3 months
* PD symptoms with evidence of stable disease as determined by the investigator
* Penile curvature deformity of >30° to <90°
* Has not had previous surgery for PD
* Has not had previous therapy with Xiaflex for PD

Exclusion Criteria:

* Ventral plaque
* Active phase PD
* Actively on anticoagulation during time frame of injections
* Aspirin 81mg will be eligible for therapy
* Hour glass deformity
* Previous allergic reaction to Xiaflex
* Unwilling to participate
* Medically unfit for sexual intercourse as deemed by the principal investigator
* Patients scheduled to undergo an elective medical procedure during the investigation timeframe that will interfere with Xiaflex injection cycles as deemed by the PI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant with previous diagnosed Peyronie's Disease will be included into the observational study at the University of Miami, Professional Art Center.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-09-02 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Psychosexual changes in Peyronie's Disease Questionnaire (PDQ). | 52 weeks
  The PDQ is highly responsive to treatment-related change in men with PD. It is self-administered, that measures psychosexual consequences after the presentation of PD. It is intended for men who have had vaginal intercourse in the past 3 months. The range of scores is from 0-24 points, with higher scores signifying greater psychosexual consequences from PD.
Penile pain evaluation in Peyronie's Disease Questionnaire (PDQ). | 52 weeks
  The PDQ is highly responsive to treatment-related change in men with PD. It measures penile pain in patients with PD. It is intended for men who have had vaginal intercourse in the past 3 months, which evaluate the levels of pain or discomfort based on last erection or vaginal intercourse. The range of scores is from 0-30 points, with higher scores signifying greater penile pain or discomfort.
Goniometer measurement to determine degree of curvature of PD. | 52 weeks
  Evaluate the total degree change of curvature improvement after treatment with Xiaflex measured by goniometer, an instrument that measures the angle of the curvature to determine the degree of the PD.

SECONDARY OUTCOMES:
International Index of Erectile Function (IIEF) Scores | 52 weeks
  The 15-question International Index of Erectile Function (IIEF) Questionnaire is a validated, multi- dimensional, self-administered investigation that has been found useful in the clinical assessment of erectile dysfunction and treatment outcomes in clinical trials. A score of 0-5 is awarded to each of the 15 questions, with a range of scores from 0-75, with lower scores signifying poorer erectile function.

CONTACTS AND LOCATIONS:
Overall Officials: Ranjith Ramasamy, MD, Principal Investigator — University of Miami
Locations (1):
- Department of Urology, University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pawlowska E, Bianek-Bodzak A. Imaging modalities and clinical assesment in men affected with Peyronie's disease. Pol J Radiol. 2011 Jul;76(3):33-7. PMID 22802839
- [Background] Levine L, Rybak J, Corder C, Farrel MR. Peyronie's disease plaque calcification--prevalence, time to identification, and development of a new grading classification. J Sex Med. 2013 Dec;10(12):3121-8. doi: 10.1111/jsm.12334. Epub 2013 Oct 4. PMID 24119147
- [Result] Gelbard M, Goldstein I, Hellstrom WJ, McMahon CG, Smith T, Tursi J, Jones N, Kaufman GJ, Carson CC 3rd. Clinical efficacy, safety and tolerability of collagenase clostridium histolyticum for the treatment of peyronie disease in 2 large double-blind, randomized, placebo controlled phase 3 studies. J Urol. 2013 Jul;190(1):199-207. doi: 10.1016/j.juro.2013.01.087. Epub 2013 Jan 31. PMID 23376148
- [Result] Lipshultz LI, Goldstein I, Seftel AD, Kaufman GJ, Smith TM, Tursi JP, Burnett AL. Clinical efficacy of collagenase Clostridium histolyticum in the treatment of Peyronie's disease by subgroup: results from two large, double-blind, randomized, placebo-controlled, phase III studies. BJU Int. 2015 Oct;116(4):650-6. doi: 10.1111/bju.13096. Epub 2015 May 18. PMID 25711400
- [Result] Kalokairinou K, Konstantinidis C, Domazou M, Kalogeropoulos T, Kosmidis P, Gekas A. US Imaging in Peyronie's Disease. J Clin Imaging Sci. 2012;2:63. doi: 10.4103/2156-7514.103053. Epub 2012 Oct 31. PMID 23230545